CLINICAL TRIAL: NCT00349284
Title: A Randomised, Double-Blind Study Comparing the Efficacy and Safety of 145 mg Fenofibrate, 10 mg Ezetimibe and Their Combination in Patients With Type IIb Dyslipidemia and Features of the Metabolic Syndrome
Brief Title: A Controlled-Study of Fenofibrate 145 mg and Ezetimibe 10 mg in Type IIb Dyslipidemic Patients With Features of the Metabolic Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C LF 178P 04 01; 2004-002408-13
Record Dates: First submitted 2006-07-05; First posted 2006-07-06 (Estimated); Last update posted 2007-09-03 (Estimated); Status verified 2007-08

CONDITIONS: Hyperlipidemia Combined
Keywords: Hyperlipidemia Combined and features of the metabolic syndrome, efficacy combination fenofibrate ezetimibe
MeSH Terms: interventions — Fenofibrate; Ezetimibe

INTERVENTIONS:
Drug: Combination of 145 mg fenofibrate and 10 mg ezetimibe

SUMMARY:
Type IIb dyslipidemia is characterized by elevated triglycerides (TG ³ 150 mg/dL), and elevated LDL-C levels (³160 mg/dL). When in addition, HDL-C is low, the presence of the lipid triad, elevated TG and LDL-C and low levels of HDL-C, seems to confer additional CHD risk in this type of patient, compared to elevated LDL-C alone.Coadministration of fenofibrate and ezetimibe could provide a complementary efficacy therapy and improve the atherogenic profile of this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Type IIb dyslipidemia.

Exclusion Criteria:

* Known hypersensitivity to fibrates or ezetimibe. Pregnant or lactating women. Contra-indication to fenofibrate or ezetimibe.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181
Dates: Start 2005-01

PRIMARY OUTCOMES:
TG and HDL-C levels.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (43):
- Belgium (16):
  - Site 113, Charleroi
  - Site 111, Comines
  - Site 112, Couillet
  - Site 115, Dessel
  - Site 114, Dour
  - Site 106, Genk
  - Site 102, Genly
  - Site 109, Kortessem
  - Site 104, Kortrijk
  - Site 108, Liège
  - Site 107, Menen
  - Site 105, Moen
  - Site 101, Oosteeklo
  - Site 110, Oostham
  - Site 116, Seraing
  - Site 103, Turnhout
- France (13):
  - Site 213, Bondy
  - Site 211, Le Beausset
  - Site 209, Nantes
  - Site 202, Orvault
  - Site 206, Paris
  - Site 208, Paris
  - Site 212, Paris
  - Site 201, Saint Sébastian Sur Loire
  - Site 205, Saint Sébastian Sur Loire
  - Site 207, Saint Sébastian Sur Loire
  - Site 203, Saint-Cyr
  - Site 210, Six-Fours-les-Plages
  - Site 204, Toulon
- Germany (14):
  - Site 313, Borna
  - Site 307, Bretten
  - Site 306, Dresden
  - Site 305, Erbach im Odenwald
  - Site 304, Frankfurt
  - Site 308, Frankfurt
  - Site 311, Frankfurt
  - Site 301, Ilvesheim
  - Site 302, Leipzig
  - Site 303, Leipzig
  - Site 314, Mannheim
  - Site 309, Offenbach
  - Site 312, Offenbach
  - Site 310, Rodgau

REFERENCES:
- [Derived] Ansquer JC, Bekaert I, Guy M, Hanefeld M, Simon A; Study Investigators. Efficacy and safety of coadministration of fenofibrate and ezetimibe compared with each as monotherapy in patients with type IIb dyslipidemia and features of the metabolic syndrome: a prospective, randomized, double-blind, three-parallel arm, multicenter, comparative study. Am J Cardiovasc Drugs. 2009;9(2):91-101. doi: 10.1007/BF03256580. PMID 19331437